CLINICAL TRIAL: NCT05211401
Title: Rituximab in Patients With ST-elevation Myocardial Infarction: A Phase 2 Placebo-controlled Randomized Clinical Trial: RITA-MI 2
Brief Title: Rituximab in Patients With ST-elevation Myocardial Infarction
Acronym: RITA-MI2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP210015; 2021-003340-24 (EudraCT Number); 2022-501893-21-00 (Other: EU Clinical Trial number)
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: ST Elevated Myocardial Infarction
Keywords: Acute Myocardial Infarction; Anterior STEMI; Rituximab; Left ventricular systolic function; CMR; Cardiac remodelling
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm 1000 mg (Experimental): Active arm 1000 mg: 1 bag containing 1000 mg of rituximab* in 500 ml of NaCl 0.9% * Mabthera® and all registered biosimilars are likely to be used in this trial.
  Interventions: Drug: Active arm 1000 mg
- Placebo arm (Placebo Comparator): 1 bag of 500 ml of NaCl 0.9%
  Interventions: Drug: Placebo arm

INTERVENTIONS:
Drug: Active arm 1000 mg — Active arm 1000 mg: 1 bag containing 1000 mg of rituximab* in 500 ml of NaCl 0.9% * Mabthera® and all registered biosimilars are likely to be used in this trial
  Arms: Active arm 1000 mg
Drug: Placebo arm — Placebo arm: 1 bag of 500 ml of NaCl 0.9%
  Arms: Placebo arm

SUMMARY:
The main objective is to compare the effect of a single injection of two doses of rituximab versus placebo on 6 months left ventricular systolic function, using CMR, in patients who have had an acute anterior STEMI. Following the sponsor's decision to stop enrolment in the 200 mg arm, the primary objective of the study is to evaluate the efficacy of a single 1000 mg dose of rituximab versus placebo.

The primary endpoint is the left ventricular ejection fraction (LVEF) by CMR at 6 months.

DETAILED DESCRIPTION:
RITA-MI 2 is an european phase IIb, multi-center, randomized, parallel, double-blind, placebo-controlled, clinical trial to assess the impact of B cell depletion with the CD20 mAb rituximab (1000mg) on left ventricular dysfunction and cardiac remodelling after acute MI.

Sample size :

372 patients, 1:1 ratio

Assessement:

Patients will be recruited immediately after admission for MI. The aim is to start the infusion of IMP within 3 hours of PPCI (defined as first balloon inflation).

Eligible patients will be offered to enter the study. In France, Spain and Czech Republic: If they accept, the investigator will collect informed written consent from the patient or from a person of trust/next of kin if the patient is unable to consent. While In Germany, UK and Netherlands, only the patient will be informed and will be able to give consent and no next-of-kin will be informed and have the possibility to give consent.

Once the inclusion is confirmed, a specific study blood sample will be taken for later assessment of cytokines and biomarkers related to immune responses, inflammation and cardiac remodelling. It will also be done at discharge and at 6 months.

According to usual practice the following blood exams will be done: Kidney function parameters (including serum creatinine, BUN, electrolytes, calcium and eGFR). It will also be done at day 5 (+ 2 days) and at 6 months.

NT-pro-BNP will be performed at admission and at 6 months. Blood leukocytes, platelets and hematologic/haemostatic parameters will also be measured at admission and at 6 months.

The randomization will be performed and the pharmacy will extemporaneously prepare (aseptically) 2 infusion bags per patient (cf. treatments below).

During the infusion, the patient will be carefully monitored with continuous cardiac telemetry:

* 12 lead ECG with QTc measurement will be performed pre-dosing and post-dosing at admission, discharge and at 6 months.
* Kidney functions. The patients will be carefully monitored by their treating physicians, as done in usual care, with a special attention to the occurrence of any adverse event related to treatment.

CMR will be done at 5 days (+ 2 days) to assess the left ventricular (LV) function, the infarct size and microvascular obstruction and at 6 months.

Study staff at the clinical sites will contact each patient at 30 days, 3 months and 12 months following randomization, by phone or during a hospital visit.

The patient participation will last after the 12-month visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with no upper limit (women must be either postmenopausal defined as being amenorrhoeic for greater than 2 years with an appropriate clinical profile, e.g. age appropriate (>55 years old), history of vasomotor symptoms) or having documented hysterectomy and/or bilateral oophorectomy) ;
* Clinical evidence at presentation of anterior ST-elevation myocardial infarction (STEMI) defined as symptoms suggestive of acute myocardial ischemia, an electrocardiogram showing ST-segment elevation ≥2 mm in ≥2 contiguous leads in V1 to V4;
* Complete occlusion (i.e. TIMI flow 0-1) of proximal or mid left anterior descending (LAD) coronary artery on urgent angiography interpreted as the infarct-related artery (IRA);
* Onset of worse symptoms within 48 hours before primary PCI;
* Patients with neutrophils >1.5 x 109/L at the moment of admission
* Patients with platelet counts >75 x 109 /L at the moment of admission
* Plan to provide primary percutaneous angioplasty (PPCI) for the patient within 2 hours of ECG diagnosis;
* Ability to start infusion of rituximab within 3 hours of PPCI ;
* Written informed consent.

Exclusion Criteria:

Exclusion Criteria :

* History of previous MI;
* Presentation with cardiac arrest;
* Cardiogenic shock (defined as systolic blood pressure <90 mmHg for >30minutes, or necessitating vasopressors to achieve a blood pressure ≥90 mmHg);
* Cardiac electrical instability (defined as complete heart block needing temporary pacing or any tachyarrhythmia needing cardioversion);
* Patients with Killip class III heart failure;
* History of severe chronic renal failure (define as stage 4 (GFR = 15-29 mL/min) or worse);
* History of hepatitis B, HIV or tuberculosis;
* Patient positive for point of care bedside test of Ag HBs;
* Severe, progressive infections documented;
* Active COVID-19 infection or COVID-19 infection within 3 months;
* Patient with documented severe immune deficiency;
* Presence, or history in ≤ five years, of an ongoing cancer, (except in situ cancer of the cervix or basal cell carcinoma);
* QTcF> 450 msecs in males, > 470msecs in females;
* Any oral or intravenous immunosuppressive treatment, immune modulatory monoclonal antibodies or immunodepleting therapy at any time (inhalers and topical creams with corticosteroids are permitted);
* Previous history of major organ transplant including renal transplant;
* Known hypersensitivity to the active substance of rituximab or to proteins of murine origin, or to any of the other excipients;
* Any contraindications to any of the rituximab premedication drugs;
* Contraindications to injectable Polaramine:

Risk of closed-angle glaucoma, Risk of urinary retention linked to urethro-prostatic disorders;

* Expected need for vaccination with a live attenuated vaccine during the study, including incomplete vaccination courses (in case, life, attenuated vaccine must be administered at least 30 days before inclusion in study);
* Absence of a complete COVID-19 vaccination scheme (including recovery from documented COVID infection) as approved at the time of enrollment in the country where the patient is recruited;
* Any obvious contraindications for MRI or conditions which will impede image acquisition for example:

Severe claustrophobia

Non-MRI compatible permanent pacemaker

Patients who have a metallic foreign body (metal silver) in their eye, or who have an aneurysm clip in their brain

Patients who have had metallic devices placed in their back

Known hypersensitivity to imaging products (gadoteric acid, meglumin or any drug containing gadolinium)

* Known hepatic failure;
* Previous history of progressive multifocal leukoencephalopathy;
* Inclusion in other interventional drug study within the previous 3 months;
* Inability to comply with study procedures;
* Patients under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) by CMR at 6 months. | 6 months
  To compare the effect of a single injection of two doses of rituximab versus placebo on 6 months left ventricular systolic function, using CMR, in patients who have had an acute anterior STEMI.

SECONDARY OUTCOMES:
Infarct size by CMR | At day 5 (+/-2) and at 6 months
  To compare the effects of rituximab versus placebo on infarct size by CMR at day 5 (+/-2) and at 6 months.
Oedema extension by CMR | At day 5 (+/-2)
  To compare the effects of rituximab versus placebo on oedema extension by CMR at day 5 (+/-2) .
T2 relaxation time at ischemic region by CMR | At day 5 (+/-2)
  To compare the effects of rituximab versus placebo on T2 relaxation time at ischemic region by CMR (using T2 mapping) at day 5 (+/-2).
Microvascular obstruction by CMR | At day 5 (+/-2)
  To compare the effects of rituximab versus placebo on microvascular obstruction by CMR (hypointense areas within LGE) at day 5 (+2/-) .
NT-pro-BNP | At 6 months
  To compare the effects of rituximab versus placebo on NT-pro-BNP at 6 months.
Adverse event related to treatment | Until 12 months
  To compare the effects of rituximab versus placebo on any adverse event related to treatment .

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel STEG, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cardiology department, Hôpital Bichat, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided